CLINICAL TRIAL: NCT06371521
Title: Ergogenic Effects of Sportlegs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Christopher Bell (Other)
Responsible Party: Sponsor-Investigator, Christopher Bell, Associate Professor, Colorado State University
Organization: Colorado State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 4933
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Performance Enhancing Product Use
Keywords: Exercise Performance; Ergogenic Aid; Lactate Supplement; Maximal Oxygen Uptake; Functional Threshold Power

STUDY DESIGN:
Intervention Model Description: Randomized, Placebo-Controlled, Double Blind Crossover Intervention
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigators and Participants are both blinded to whether the participants will be consuming Sportlegs or Placebo during a given study visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VO2max and Lactate Threshold (Experimental): Participants will ingest either Sportlegs or placebo.
  The Sportlegs (and placebo) will be ingested as dietary capsules taken with water.
  30-minutes after ingestion, the VO2max and lactate threshold testing will commence. This will involve a graded exercise test on a cycle ergometer to volitional fatigue. Heart rate and gas exchange will be measured prior to and throughout the exercise test. Blood will be sampled approximately every 60-seconds from a venous catheter placed in a hand or wrist vein, or from a finger using a lancet and cappillary tube. The amount of blood to be sampled is up to ~2-3 ml per sample, totalling less than 40 mL per lab visit. The blood will be immediately analyzed for lactate concentration using an automated analyzer. Ratings of Perceived Exertion will be recorded every ~2 minutes.
  VO2max and lactate threshold are considered important predictors of exercise performance.
  Interventions: Dietary Supplement: Sportlegs; Dietary Supplement: Placebo
- Maximal Mean Power Output (Experimental): The Sportlegs (and placebo) will be ingested as dietary capsules taken with water.
  30-minutes after ingestion, participants will begin the FTP20 test. Following a brief, standardized warm-up, participants will exercise on a stationary cycle ergometer at the highest intensity they are able to sustain for 20-minutes. This is akin to a "time-trial" where cyclists cover as greater distance as possible during a pre-determined period of time. During the FTP20 test, work rate will be monitored and recorded, as will heart rate (monitored continuously but only recorded every 5-minutes via short range telemetry or ECG). Rating of perceived exertion will also be assessed and recorded every 5-minutes.
  The FTP20 test is considered an important predictor of exercise performance.
  Interventions: Dietary Supplement: Sportlegs; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Sportlegs — Sportlegs contains lactate (from calcium lactate pentahydrate and magnesium lactate dihydrate), magnesium (from magnesium lactate dihydrate), calcium (from calcium lactate pentahydrate), and vitamin D (as cholecalciferol).
Dietary Supplement: Placebo — Empty Capsules to serve as a placebo control

SUMMARY:
Sportlegs is a commercially available dietary/sports supplement. It is manufactured by a local, Colorado-based company: Sport Specifics Inc. Although Sportlegs has been on the market for approximately 20-years, very little empirical research has been completed to determine if Sportlegs improves exercise performance. Sport Specifics Inc. has commissioned Colorado State University to investigate the ergogenic effects of Sportlegs.

DETAILED DESCRIPTION:
1. Study Significance: Based on published survey data, it is estimated that more than 50% of Americans consume dietary supplements, including sport drinks. In light of widespread use, research that evaluates the claims made by the manufacturers of supplements and sport drinks appears to be relevant to a great number of people. Scientific evaluation of Sportlegs will provide potential customers with an opportunity to make an informed decision as to how they wish to spend their money.
2. Sport Specifics Inc., has had considerable commercial success selling their product, Sportlegs. However, they recognize the potential benefit of being able to support claims pertaining to the efficacy of their product with peer-reviewed scientific data. Noteworthy, they also are aware of the potential risks of a scientific evaluation that may demonstrate that their product has no effect on exercise performance, or possibly even a negative/unfavorable effect.
3. Literature Review: To date, only one scientific study of Sportlegs has been published (see attached). The data suggest that Sportlegs may increase blood bicarbonate concentration (an important factor controlling blood pH) and fatigue resistance, as described by time to exhaustion.
4. The primary ingredient in Sportlegs is lactate. Lactate is a modified form of sugar (glucose) and is therefore a potentially important source of fuel for exercise. In this regard, the potential for Sportlegs to improve exercise performance by making more fuel available is intuitively appealing.
5. Historical thinking has misclassified lactic acid as metabolic waste product, and a potential source of fatigue and muscle damage. The modern contemporary opinion is that lactate is a gluconeogenic precursor (i.e. a source of glucose), an excellent source of chemical energy for many organs including the heart and skeletal muscle, and it may even have favorable clinical relevance with respect to a number of chronic diseases (see attached review for more details). The current proposed work may contribute to the field of Exercise Physiology by providing further confirmation of the functional benefits of lactate and correcting previously erroneous interpretations of data.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30 years (inclusive)
* Minimum of 150 minutes/week of moderate intensity endurance exercise during the previous 12-months.

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Use of Sportlegs within the previous 4-weeks
* Use of magnesium supplements within the previous 4-weeks
* Unwillingness to abstain from the use of other potentially ergogenic dietary supplements throughout the duration of participation in the study
* Inability or unwillingness to perform vigorous cycle ergometer exercise

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Maximal Oxygen Uptake | 30 minutes following Sportlegs or Placebo ingestion.
  To compare VO2max, determined during incremental stationary cycle ergometer exercise, in young healthy adults after acute ingestion of placebo and Sportlegs.
Lactate Threshold | 30 minutes following Sportlegs or Placebo ingestion
  To compare lactate threshold, determined during incremental stationary cycle ergometer exercise, in young healthy adults after acute ingestion of placebo and Sportlegs.
Rating of Perceived Exertion (RPE) | During the VO2max and maximal mean power tests
  To compare perceived rates of exertion, determined during stationary cycle ergometer exercise, in young healthy adults after acute ingestion of placebo and Sportlegs.
Maximal sustained mean power | 30 minutes following Sportlegs or Placebo ingestion
  To compare the maximal mean power that can be sustained on a cycle ergometer for 20-min, in young healthy adults after acute ingestion of placebo and Sportlegs.

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No